CLINICAL TRIAL: NCT00280982
Title: Vaccination With Autologous Dendritic Cells Pulsed With Tumor Lysate for Treatment of Patients With Malignant Pleural Mesothelioma
Brief Title: Dendritic Cell-based Immunotherapy in Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Erasmus MC, Pulmonary Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2005-269; PMR-MM05-001
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: dendritic cells, immunotherapy, vaccination, mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma

INTERVENTIONS:
Biological: tumor lysate-loaded autologous dendritic cells — 50x10e6 cells per vaccination, 3 times, 2 weeks interval
  Other Names: DC

SUMMARY:
Exploiting the immunostimulatory capacities of dendritic cells holds great promise for cancer immunotherapy. A mouse model for malignant mesothelioma allowed us to prove that autologous dendritic cells presenting tumor antigens were very effective by (partly) inhibiting tumor growth. This study will test the feasibility and safety of a clinical trial using autologous DC as a therapeutic adjuvant for the treatment of malignant pleural mesothelioma.

DETAILED DESCRIPTION:
For this phase I study, patients with end-stage malignant mesothelioma and who are deemed to be fit enough to be treated with chemotherapy will be asked to participate in this study. Patients will first be treated with 4 courses of chemotherapy (standard treatment[Alimta/cisplatin]). After this chemotherapy a leukapherese is performed of which the monocytes are used for differentiation to dendritic cells. The procedure to grow these dendritic cells in vitro (culture) and pulse them with tumor lysate is performed in a cleanroom environment. Several quality control tests will be performed before the dendritic cells are ready for re-injection. Three doses of properly pulsed autologous dendritic cells are then re-injected every two weeks.

Using the proper procedure in mesothelioma patients, minor side effects are expected.

Ten (10) patients will be treated by this procedure to define the safety and toxicity of immunization and to observe (anti-tumor) immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically and histological or cytological confirmed newly diagnosed mesothelioma, that can be measured in two dimensions by a radiologic imaging study.
* Patients must be at least 18 years old and must be able to give written informed consent.
* Patients must be ambulatory (Karnofsky scale > 70, or WHO-ECOG performance status 0,1, or 2) and in stable medical condition. The expected survival must be at least 4 months.
* Patients must have normal organ function and adequate bone marrow reserve: absolute neutrophil count > 1.5*109/l, platelet count > 100*109/l, and Hb > 6.0 mmol/l.
* Positive delayed type hypersensitivity skin test (induration > 2mm after 48hrs) against at least one positive control antigen of MULTITEST CMI (Pasteur merieux).
* Stable disease or response after chemotherapy.
* Availability of sufficient tumor material of the patient.
* Ability to return to the Erasmus MC for adequate follow-up as required by this protocol.

Exclusion Criteria:

* Conditions that make the patient unfit for chemotherapy or progressive disease after 4 cycles of chemotherapy.
* Pleurodesis at the affected side before the pleural fluid is obtained.
* Medical or psychological impediment to probable compliance with the protocol.
* Patients on steroid (or other immunosuppressive agents) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation and must stop of any such treatment during the time of the study.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, superficial or in-situ cancer of the bladder or other cancer for which the patient has been disease-free for five years.
* Serious concomitant disease, no active infections. Patients with a history of autoimmune disease or organ allografts, or with active acute or chronic infection, including HIV and viral hepatitis.
* Patients with serious intercurrent chronic or acute illness such as pulmonary (asthma or COPD) or cardiac (NYHA class III or IV) or hepatic disease or other illness considered by the study coordinators to constitute an unwarranted high risk for investigational DC treatment.
* Patients with a known allergy to shell fish (contains KLH).
* Pregnant or lactating women.
* Patients with inadequate peripheral vein access to perform leukapheresis
* Concomitant participation in another clinical trial
* An organic brain syndrome or other significant psychiatric abnormality which would comprise the ability to give informed consent, and preclude participation in the full protocol and follow-up.
* Absence of assurance of compliance with the protocol. Lack of availability for follow-up assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
safety | april 2008
tolerability | april 2008

CONTACTS AND LOCATIONS:
Overall Officials: Joachim G Aerts, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Department of Pulmonary Medicine, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Hegmans JP, Hemmes A, Aerts JG, Hoogsteden HC, Lambrecht BN. Immunotherapy of murine malignant mesothelioma using tumor lysate-pulsed dendritic cells. Am J Respir Crit Care Med. 2005 May 15;171(10):1168-77. doi: 10.1164/rccm.200501-057OC. Epub 2005 Mar 11. PMID 15764728
- [Derived] Hegmans JP, Veltman JD, Lambers ME, de Vries IJ, Figdor CG, Hendriks RW, Hoogsteden HC, Lambrecht BN, Aerts JG. Consolidative dendritic cell-based immunotherapy elicits cytotoxicity against malignant mesothelioma. Am J Respir Crit Care Med. 2010 Jun 15;181(12):1383-90. doi: 10.1164/rccm.200909-1465OC. Epub 2010 Feb 18. PMID 20167848